CLINICAL TRIAL: NCT04938401
Title: Construction and Application of a Risk Prediction Model Forepistaxis After Endoscopic Transsphenoidal Pituitary Tumor Resection
Brief Title: Construction and Application of a Risk Prediction Model Forepistaxis After Pituitary Tumor Resection
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Wang Ying supervisor nurse (Other)
Collaborators: Sir Run Run Shaw Hospital (Other); Zhejiang University (Other); Zhejiang Provincial People's Hospital (Other)
Responsible Party: Sponsor-Investigator, Wang Ying supervisor nurse, Neurosurgery 5 Ward, Second Affiliated Hospital, School of Medicine, Zhejiang University
Organization: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Other Study IDs: Neurosurgery 5 Ward
Record Dates: First submitted 2021-06-01; First posted 2021-06-24 (Actual); Last update posted 2021-06-24 (Actual); Status verified 2021-06

CONDITIONS: Pituitary Tumor
MeSH Terms: conditions — Pituitary Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: US Export: No

GROUPS / COHORTS (2):
- epistaxis: Postoperative pituitary tumor group with epistaxis
- no epistaxis: Postoperative pituitary tumor group without epistaxis

INTERVENTIONS:
Other:

SUMMARY:
(1) Objective to establish an evaluation system for predicting the risk of epistaxis after endoscopic transsphenoidal pituitary surgery（ 2) Objective to determine the risk factors of epistaxis after endoscopic transsphenoidal pituitary adenoma surgery. Referring to domestic and foreign literature, combined with experts' opinions, the related risk factors that may cause postoperative nosebleed of pituitary adenoma are: 22 patients and surgical factors. 3) Objective to establish a risk prediction model of epistaxis after endoscopic transsphenoidal pituitary tumor resection. According to the occurrence of epistaxis, the patients in the modeling group were divided into epistaxis group and non epistaxis group. The risk factors of epistaxis were taken as the independent variable, and the occurrence of epistaxis was taken as the dependent variable. The variables with statistical significance in univariate analysis were included in the multivariate logistic regression model, and the risk prediction model of epistaxis after pituitary tumor resection was established by back LR method.(4) Objective to verify the risk prediction model of endoscopic transsphenoidal pituitary adenoma epistaxis. The validation model is used to validate the prediction model, and the Hosmer-Lemeshow degree is used to match the model. The area under the receiver operating characteristic curve (ROC) was used to evaluate the validity of the model.(5) Application of risk prediction model.

ELIGIBILITY:
Inclusion Criteria:

Those who met the diagnostic criteria of pituitary tumor and received transsphenoidal endoscopic surgery during hospitalization; Patients with informed consent; Age ≥ 14 years old.

Exclusion Criteria:

quitters; patients with incomplete clinical data;

Ages: 14 Years to 90 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients after transnasal sphenoidal resection of pituitary tumor
Sampling Method: Non-Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2021-07-02 (Estimated); Primary Completion 2021-10-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of epistaxis | up to 24 weeks
  Overall incidence of epistaxis

CONTACTS AND LOCATIONS:
Overall Officials: YIing Wang, Study Chair — Second Affiliated Hospital, School of Medicine, Zhejiang University

IPD SHARING:
Plan to Share IPD: Undecided